CLINICAL TRIAL: NCT07244432
Title: Post-ERCP Pancreatitis- Prophylactic Measures Implementation Study
Brief Title: Post-ERCP Pancreatitis - Prophylactic Measures Implementation Study (PEP-PROMIS)
Acronym: PEP-PROMIS
Status: Not yet recruiting | Type: Observational
Sponsor: Branislav Kuncak (Other)
Responsible Party: Sponsor-Investigator, Branislav Kuncak, Head of Gastroenterology, Principal Investigator, MD, University Hospital Bratislava
Organization: University Hospital Bratislava (Other)
Other Study IDs: NSM-BA-PEP-PROMIS
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Pancreatitis, Acute; ERCP; Prophylaxis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consecutive adult patients with native papilla undergoing ERCP at participating centers.: Consecutive adult patients undergoing first endoscopic retrograde cholangiopancreatography (ERCP) or repeat ERCP after a previous failed cannulation attempt who have provided signed informed consent will be included. Patients will be excluded if they have a history of papillotomy, papilla dilation, or sphincteroplasty; if the rendezvous cannulation technique is used; if they show insufficient cooperation preventing cannulation; or if the ERCP is terminated before cannulation due to sedation- or anesthesia-related complications. Additional exclusion criteria include failure to reach the major or minor papilla (for example, due to duodenal stenosis), acute biliary pancreatitis, or altered anatomy preventing access to the papilla with a standard duodenoscope (such as Roux-en-Y reconstruction). The standard ERCP procedure will be performed under analgosedation or general anesthesia, depending on the patient's condition and the institutional protocol.

SUMMARY:
This is a prospective, observational (non-interventional), multicenter study that will look at how often inflammation of the pancreas (called post-ERCP pancreatitis, or PEP) occurs after an endoscopic procedure known as ERCP. The study will take place in several hospitals in Slovakia and Czechia and will include all patients who have this procedure during the study period.

ERCP is a common procedure used to treat problems in the bile ducts and pancreas. Although generally safe, it sometimes leads to PEP, which is the most frequent and potentially serious complication. Monitoring the rate of PEP helps doctors evaluate the overall quality of ERCP procedures, since patient safety is an important part of quality care.

The study will also look at how well hospitals follow current prevention guidelines from two major professional organizations-the European Society of Gastrointestinal Endoscopy (ESGE) and the American Society for Gastrointestinal Endoscopy (ASGE)-and how these prevention methods affect the risk of PEP. This information will help identify how closely real-world practice follows recommended preventive measures and provide new data about PEP rates in the region.

ELIGIBILITY:
Inclusion Criteria:

* ERCP in a patient with a native papilla (first ERCP) or repeat ERCP in a patient with previous failed cannulation attempt.
* Age at least 18 years at the time of ERCP.
* Signed informed consent.

Exclusion Criteria:

* Previous papillotomy, papilla dilation, or sphincteroplasty.
* Rendez-vous cannulation technique.
* ERCP not performed due to insufficient patient cooperation.
* ERCP terminated before cannulation due to sedation/anesthesia-related complications.
* Failure to reach the Vater's or minor papilla (e.g. duodenal stenosis).
* Acute biliary pancreatitis.
* Altered anatomy that prevents reaching the papilla with a standard duodenoscope (e.g. Roux-en-Y).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adults undergoing ERCP at participating centers. Selected ERCP centers within the Slovakia and Czechia. The centers selected for this study are those that expressed interest in participating based on our yet unpublished 2024 survey, which aimed to assess how ERCP quality parameters were monitored and how prophylactic measures for PEP were implemented across centers. A total of 26 ERCP centers participated in the survey, including 14 from Slovakia and 12 from Czechia. Centers that expressed interest, as well as all remaining ERCP-performing centers in Slovakia and several in Czechia, were subsequently contacted by email with information about the study and invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who develop post-ERCP pancreatitis. | 48 hours after the procedure.

SECONDARY OUTCOMES:
Percentage of participants experiencing none, mild, moderate, or severe post-ERCP pancreatitis. | Every 7 days until hospital discharge.
Proportion of ERCP procedures in which one or more guideline-recommended preventive measures are used. | Periprocedural preventive measures applied immediately before, during, or shortly after the ERCP procedure. Aggressive hydration may continue for up to 8 hours post-procedure.
Number of participants stratified by predefined patient- and procedure-related risk factors and occurrence of post-ERCP pancreatitis | Periprocedurally
  Includes age, sex, ERCP indication, and ESGE-defined patient- and procedure-related risk factors
Number of participants with PEP-related mortality during index hospitalization or within 30 days after ERCP. | Up to 30 days post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Martinek, Prof, MD, Ph.D, Study Chair — Gastroenterology, St. Anne´s University Hospital, Brno, Czech Republic; Branislav Kunčak, MUDr., Principal Investigator — St. Michael´s University Hospital and Slovak Health University, Bratislava, Slovakia

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-11-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT07244432/SAP_000.pdf